CLINICAL TRIAL: NCT04916964
Title: Effects of the Adapted Home-based Exercise Program "T&E" (Test-and-Exercise) on Balance, Mobility, and Executive Functions in Persons With Alzheimer's Disease: Protocol for an Exploratory Pilot Study
Brief Title: Adapted Home-based Exercise Program "T&E" (Test-and-Exercise) in Persons With Alzheimer's Disease (HOPE Trial)
Acronym: HOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HES-SO Valais-Wallis (Other)
Collaborators: Hilfiker Roger (Unknown)
Responsible Party: Principal Investigator, Mittaz Hager Anne-Gabrielle, Professor, HES-SO Valais-Wallis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOPE
Record Dates: First submitted 2021-05-31; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Home-based exercise program; Basic functional mobility; Central executive functions
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test & Exercise home-based program (T&E) (Experimental): Eight home-based physiotherapy sessions will occur in two months, once a week
  Interventions: Other: Test and exercise home-based program

INTERVENTIONS:
Other: Test and exercise home-based program — Eight home-based physiotherapy sessions will occur in two months, once a week, to activate the preserved implicit memory (PIM). The recommendations are to train three weeks with the same exercise program, three times a week (one time coached by the attributed physiotherapist and two times coached by a natural or family caregiver). After three weeks, the participants can choose if they want to keep the same exercises or change all or some of these, in testing other tasks. Every training session will be planned to last 45 minutes. During each training session, the participant will note on his/her own "Training booklet" each task performed. The "Training booklet" will be used to plane, organize, and remember details for the next training session.
  Other Names: T&E

SUMMARY:
The aim of this exploratory pilot study is to assess the feasibility and effectiveness of the adapted T&E home-based exercise program on the basic functional mobility and executive functions in persons with mild or probable Alzheimer's Disease.

DETAILED DESCRIPTION:
Primary and secondary outcomes will be measured at T0 (one week before the begin of the intervention) and T1, (one week after the eight weeks of the intervention) at home of the participants.

Eight home-based physiotherapy sessions will occur in two months, once a week, to activate the preserved implicit memory (PIM). The recommendations are to train three weeks with the same exercise program, three times a week (one time coached by the attributed physiotherapist and two times coached by a natural or family caregiver). After three weeks, the participants can choose if they want to keep the same exercises or change all or some of these, in testing other tasks. Every training session will be planned to last 45 minutes. During each training session, the participant will note on his/her own "Training booklet" each task performed. The "Training booklet" will be used to plane, organize, and remember details for the next training session.

Twelve participants will take part at this study.

ELIGIBILITY:
Inclusion Criteria:

* Must living at their own home,
* Clinical diagnosis of mild or probable Alzheimer's Disease,
* Must be medical stable,
* Must be able to walk with or without assistive device without physical assistance of another person,
* Must be able to follow one-step commands,
* Family caregiver's must agree to participate at the training sessions.

Exclusion Criteria:

* Severe vision and verbal impairment,
* Any serious orthopaedic condition,
* Any major neurologic or musculoskeletal comorbidity that might affect their functional mobility,
* Any limiting cardiac or pulmonary condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional mobility | 8 weeks
  Berg Balance Scale (BBS), scoring ranges from 0 (worse) to 56 (best)
Stand and go | 8 weeks
  Time Up and Go test (TUG) in seconds
Sit to stand | 8 weeks
  Five Time Sit to Stand (FTSTS) in seconds
Walking speed | 8 weeks
  The self-selected and the maximal walking speed (SSWS/MWS) on a 6-meter walk

SECONDARY OUTCOMES:
The Set shifting (Mental flexibility) | 8 weeks
  Trail Making Test Part-Be in seconds
The updating (Working memory) | 8 weeks
  Digit span backward task, number of the successful sequences between 0 and 14
The response inhibition | 8 weeks
  Stroop Color and Word Test (SCWT) Victoria, comparison of the expected score to the participant's score to calculate the Z-score
Feasibility of recruitement | 4 months
  Inclusion of 12 subjects between the 30 of May 2021 ant the 30 of Septembre 2021
Participation agreement | 4 months
  Fulfilled if 75% of eligible subjects agree to participate and sign the consent
Costs | 8 months
  Fulfilled if the cost does not exceed the planed amounts by more than 5%
Drop out / withdraw | 8 months
  Fulfilled if 75% of the participants take part in the total duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Gabrielle Mittaz Hager, PhD Cand, Principal Investigator — HES-SO Valais-Wallis
Locations (1):
- CMS Sierre Région, Sierre, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrard S, Eyer S, Hilfiker R, Mittaz Hager AG. Adapted Home-Based Exercises in Dementia: An Exploratory Pre-post Pilot and Feasibility Study. Am J Alzheimers Dis Other Demen. 2024 Jan-Dec;39:15333175241263741. doi: 10.1177/15333175241263741. PMID 38877608